CLINICAL TRIAL: NCT03138902
Title: Validation of Carbohydrate Intolerance Questionnaire
Brief Title: Carbohydrate Intolerance Questionnaire Study
Acronym: Curves1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Curves International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2013-0401
Record Dates: First submitted 2017-04-25; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Carbohydrate Intolerance
MeSH Terms: conditions — Glucose-Galactose Malabsorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glucose Tolerance Beverage (Experimental): 75 g. of a fruit punch flavored oral glucose solution
  Interventions: Dietary Supplement: TRUTOL Glucose Tolerance Beverage

INTERVENTIONS:
Dietary Supplement: TRUTOL Glucose Tolerance Beverage — A caffeine-free, non-carbonated, glucose tolerance beverage

SUMMARY:
The purpose of this study is to evaluate the validity of using a carbohydrate intolerance questionnaire (CIQ) and/or other health markers as a means of predicting response to insulin sensitivity as determined by an oral glucose tolerance test (OGTT).

DETAILED DESCRIPTION:
This study will utilize a carbohydrate intolerance questionnaire (CIQ). Responses to a CIQ will be correlated with diet inventories, baseline body composition and health assessments, a standard metabolic panel, fasting glucose and insulin levels, a homeostatic insulin resistance model (HOMA), a two hour oral glucose tolerance test (OGTT), and a carbohydrate sensitivity symptom questionnaire administered during the OGTT.

ELIGIBILITY:
Inclusion Criteria:

* Participant is female
* Participant is between the ages of 18 and 60

Exclusion Criteria:

* Participant is pregnant or nursing
* Participant is diabetic or pre-diabetic
* Participant has a Body Mass Index (BMI) < 22

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females were requested by the Sponsor
Enrollment: 108 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Complete a Carbohydrate Intolerance Questionnaire (CIQ) | 1 day
  Primary Outcome
Complete a 2 Hour Oral Glucose Tolerance Test (OGTT) to measure glucose response | 2 hours
  Primary Outcome
Complete a 2 Hour Oral Glucose Tolerance Test (OGTT) to measure insulin response | 2 hours
  Primary Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No